CLINICAL TRIAL: NCT06512467
Title: Donafenib Combine With Sintilimab and HAIC in Neoadjuvant of Resectable Hepatocellular Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20240499
Record Dates: First submitted 2024-07-16; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular Carcinoma; Donafenib; Sintilimab; HAIC
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib; sintilimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donafenib combined with Sintilimab and HAIC (Experimental): Donafenib:200mg bid; Sintilimab:200mg Q3D; HAIC:Q3W.
  Interventions: Drug: Donafenib; Drug: Sintilimab; Other: HAIC

INTERVENTIONS:
Drug: Donafenib — 200 mg BID,oral administration will start before the first HAIC treatment .
Drug: Sintilimab — 200 mg Q3W,Intravenous infusion will perform before HAIC treatment.
Other: HAIC — HAIC,Q3W. The total number of HAIC treatments was determined by the investigator based on patient needs. Dose: Oxaliplatin 85 mg / m2 for 2h, Calcium folinate 400 mg / m2 for 2h, 5-FU 400 mg / m2 for 10min, followed by 5-FU 1200 mg / m2 for 23 hours).

SUMMARY:
The investigators design a phase IIB clinical study to explore the efficacy and safety of Donafenib combined with Sintilimab and HAIC in neoadjuvant of resectable Hepatocellular Carcinoma.

DETAILED DESCRIPTION:
This trial is a single-arm, non-randomized and single-center clinical study of Donafenib combined with Sintilimab and HAIC in Neoadjuvant of Resectable Hepatocellular CarcinomaIt will estimate that 30 patients who met the study criteria will be enrolled in Tianjin Medical University Cancer Institute and Hospital and neoadjuvant in Donafenib combined with Sintilimab and HAIC. The investigators will follow up and collect subjects' data monthly to evaluate the efficacy and safety of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily join the study and sign the informed consent;
2. Age 18 ~ 80 years old (including 80 years old), male and female;
3. Patients with hepatohcellular carcinoma diagnosed clinically or confirmed by histology / cytology according to the code for diagnosis and treatment of primary liver cancer (2022 Edition);
4. Hepatocellular carcinoma and technically resectable (CNLC stage Ⅱb to Ⅲa), estimated residual liver volume >30%, in patients with cirrhosis, the residual liver volume is >40%. And meets at least one of the following conditions:

   1. The tumor is adjacent to large blood vessels or other organs, resulting in an expected surgical margin of less than 1cm;
   2. Cancer thrombus formation was associated with ipsilateral portal vein or hepatic vein, but the tumor thrombus did not accumulate in the main contralateral portal vein, contralateral portal vein, contralateral hepatic vein, and superior mesenteric vein;
5. At least one assessable lesion (mRECIST criteria),and did not receive radiotherapy or local treatmen;
6. ECOG 0 ~ 1;
7. Major organs are functioning normally. Hemoglobin ≥ 90 g / L; ANC ≥ 1.5 × 109/L； Platelet count ≥ 100 × 109/L； Albumin ≥ 28 g / L; Total bilirubin ≤ 3 × ULN; AST, ALT ≤ 5 × ULN； TSH ≤ ULN； INR or PT ≤ 1.5 × ULN, APTT ≤ ULN.
8. If HBsAg (+) and/or anti-HCV (+), antiviral therapy should be standard based on HBV DNA or HCV RNA test results;
9. Be able to cooperate to observe adverse events. -

Exclusion Criteria:

1. Cholangiocarcinoma, mixed cell carcinoma and fibrous laminar cell carcinoma are known
2. Diffuse tumor lesions
3. extrahepatic metastasis
4. Active malignancies other than HCC occur within 5 years or at the same time, with the exception of cured skin basal cell carcinoma, cervical carcinoma in situ and thyroid form carcinoma;
5. Received radical hepatectomy, systemic anticancer therapy for liver cancer (mainly including systemic chemotherapy, molecular targeted therapy, CTLA-4, PD-1/PD-L1 monoclonal antibody immunotherapy) and local liver therapy, including TACE, HAIC, TAE, local ablation, radiotherapy, etc;
6. The following conditions were present during the course of the study: myocardial infarction, severe unstable angina pectoris, NYHA2 or higher cardiac insufficiency, poor arrhythmia control, symptomatic congestive heart failure, cerebrovascular accident;
7. A history of hypertensive crisis or hypertensive encephalopathy;
8. The subject has any history of active autoimmune disease or autoimmune disease (but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitaritis, vasculitis, nephritis, hyperthyroidism, hypothyroidism; Subjects with vitiligo or childhood asthma are in complete remission and can be included as adults without any intervention; Asthma requiring medical intervention with bronchodilators will not be included);
9. Subjects are receiving immunosuppressive, systemic or absorbable local hormone therapy for immunosuppressive purposes and continue to receive such therapy during the 2 weeks prior to enrollment;
10. Abnormal coagulation (INR > 1.5 or APTT > 1.5 x ULN) with bleeding tendency or receiving thrombolysis or anticoagulation therapy;
11. Known severe adverse reactions to Donafenib, sindillizumab, or severe allergic reactions to other monoclonal antibodies;
12. The subject has a known history of psychotropic, alcohol, or drug abuse. -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
MPR(Major Pathological Response) | 1 year
  After neoadjuvant therapy, the proportion of residual tumor cells was less than 30%.

SECONDARY OUTCOMES:
ORR(Objective Response Rate) | 1 year
  The rate of participants that achieve either a complete response (CR) or a partial response (PR).
DCR(Disease Control Rate) | 3 year
  The percentage of cases with remission (PR + CR) and stable lesions (SD) after treatment was assessable.
RFS(Recurrence-free Survival) | 1 year
  The time experienced from the enrollment date until tumor recurrence or death from any cause, if the subject died before the disease recurred. Survival subjects whose tumor recurrence was not confirmed by the database deadline were deleted according to the date of the last imaging tumor assessment. The date of tumor recurrence was the date of the first imaging confirmation of tumor recurrence.
OS(Overall Survival) | 3 year
  Overall survival is defined as time from the start of treatment until death due to any reason.
  R0 resection： The tumor was completely resected, and the submicroscopic margin was negative, that is, no tumor remained.
pCR(Pathological Complete Response) | 1 year
  No residual tumor was found pathologically in patients with neoadjuvant therapy induced tumor regression.